CLINICAL TRIAL: NCT00242437
Title: A Prospective, Multicenter Study to Evaluate Hemostatic Matrix With Bovine Thrombin in Achieving Hemostasis in Patients Undergoing Endoscopic Sinus Surgery
Brief Title: Hemostatic Matrix in Endoscopic Sinus Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 400-05-002
Record Dates: First submitted 2005-10-19; First posted 2005-10-20 (Estimated); Last update posted 2006-07-13 (Estimated); Status verified 2006-07

CONDITIONS: Sinusitis
MeSH Terms: conditions — Sinusitis

INTERVENTIONS:
Device: Hemostatic matrix
Device: bovine thrombin

SUMMARY:
Evaluating clinical performance of Hemostatic Matrix with bovine thrombin in achieving hemostasis in patients undergoing endoscopic sinus surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years or older.
* Patients undergoing elective primary or re-do endoscopic sinus surgery for chronic sinusitis with bleeding surface requiring an adjunct to achieve hemostasis.
* Patients must be willing and capable of cooperating to the extent and degree required by the protocol and sign the IRB approved Informed Consent Form prior to any participation in the study.

Exclusion Criteria:

* Patients with bleeding diathesis, pathologic coagulopathy, systemic disorders, inflammatory conditions (other than chronic sinusitis or nasal polyposis) or autoimmune, immunodeficiency diseases or any other disorder that may interfere with hemostasis.
* Patients with severe (brisk or forceful) bleeding site(s).
* Patients undergoing urgent or emergency endoscopic sinus surgery.
* Patients with bronchial asthma who have aspirin intolerance.
* Patients with diffuse polyposis that would require chronic oral steroids or patients on chemotherapeutic agents that might delay healing (short term pulse steroid therapy and topical steroids are acceptable).
* Patients who have used anticoagulant, antiplatelet or nonsteroidal anti-inflammatory analgesic (NSAID) within 7 days prior to surgery.
* Patients who are morbidly obese (Body Mass Index > 35).
* Patients with acute local infection at the operative side.
* Patients who are current alcohol and/or drug abusers.
* Patients with neoplasm, craniofacial abnormalities (e.g. cleft palate), or sleep apnea using nasal CPAP, or patients that may require a Lothrop procedure.
* Female patients who are pregnant or nursing.
* Patients who have uncontrolled diabetes mellitus (blood glucose levels >400 mg/dl) as determined by the Investigator based on medical history.
* Patients who have participated in another investigational drug or device research within 30 days of enrollment.
* Patients with known antibodies to bovine thrombin preparations, sensitivities or religious prohibitions to porcine gelatin or bovine components.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-10; Study Completion 2006-02

PRIMARY OUTCOMES:
Success in achieving hemostasis after product application

SECONDARY OUTCOMES:
Post operative healing
Patient Satisfaction
Time to hemostasis

CONTACTS AND LOCATIONS:
Overall Officials: James Hart, MD, Study Director — Ethicon, Inc.
Locations (3):
- United States (3):
  - The Summit Medical GroupDepartment of Otolaryngology, Summit, New Jersey
  - The Medical University of South Carolina Department of Otolaryngology, Charleston, South Carolina
  - University of Tennessee Department of Otolaryngology, Memphis, Tennessee